CLINICAL TRIAL: NCT03906942
Title: Using Team Science to Promote Health-Enhancing Physical Activity in Adults With Obesity in a Community Setting: A Feasibility Study
Brief Title: Team Science to Promote Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: University of Miami (Other); Sparrow Health System (Other)
Responsible Party: Principal Investigator, Nicholas Myers, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: STUDY00002012
Record Dates: First submitted 2019-04-03; First posted 2019-04-08 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Health Promotion
MeSH Terms: interventions — Health

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the Fun For Wellness (FFW) group or the Usual Care (i.e., UC) group by the code programmed within the FFW website that is specified to achieve a 1:1 group (i.e., nFFW = 15, nUC = 15) assignment. Participants assigned to the UC group (i.e., UC participants) will proceed through the pre-operative weight management program provided by the center. Participants assigned to the FFW group (i.e., FFW participants) will proceed through the pre-operative program provided by the center and will be given 4 weeks (i.e., Week 3 through Week 6) of 24 hr access to the FFW online intervention during data collection for this study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, center staff, and research staff will be blinded to participant group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fun For Wellness (FFW) (Experimental): Participants assigned to the FFW group (i.e., FFW participants) will proceed through the pre-operative program provided by the center and will be given 4 weeks of 24 hr access to the FFW online intervention during data collection for this study. Intervention participants will: 1) watch original videos with vignettes performed by professional actors; 2) read and/or watch mini-lectures that teach skills for behavior change; 3) engage in self-reflection exercises, 4) play original interactive games related to vignettes and mini-lectures; 5) interact with other FFW users via chat room functions and; 6) watch funny narrated video clips about well-being and/or physical activity.
  Interventions: Behavioral: Fun For Wellness (FFW)
- Usual Care (UC) (No Intervention): Participants assigned to the UC group (i.e., UC participants) will proceed through the pre-operative weight management program provided by the center.

INTERVENTIONS:
Behavioral: Fun For Wellness (FFW) — FFW consists of videos, games, and content in the form of 152 BET I CAN challenges [1]. Behavior challenges are intended to increase a participant's capabilities to set a goal and to create positive habits. Emotion challenges are intended to increase a participant's capabilities to cope with negative emotions and to cultivate positive emotions. Thought challenges are intended to increase a participant's capabilities to challenge negative assumptions and to create a new narrative for their life. Interaction challenges are intended to increase a participant's capabilities to communicate and connect with others. Context challenges are intended to increase a participant's capabilities to read cues and to change cues in the environment. Awareness challenges are intended to increase a participant's capabilities to know herself/himself and to know the issue. Next steps challenges are intended to increase a participant's capabilities to make a plan and to stick with a plan.
  Arms: Fun For Wellness (FFW)

SUMMARY:
Background: Fun For Wellness is an online intervention designed to promote growth in well-being and physical activity by providing confidence-enhancing learning opportunities to participants.

Objective: The objective of this feasibility study is to address uncertainties regarding the inclusion of accelerometer-based assessment of physical activity within the Fun For Wellness online intervention among free-living adults with obesity in the United States of America.

Method: The study design is a prospective, double-blind, parallel group randomized pilot trial.

Discussion: Results are intended to inform the preparation of a future definitive randomized controlled trial.

DETAILED DESCRIPTION:
Fun For Wellness is an online intervention designed to promote growth in well-being and physical activity by providing confidence-enhancing learning opportunities to participants [1]. The conceptual framework for the Fun For Wellness intervention is guided by self-efficacy theory [2]. Evidence has been provided for the efficacy of Fun For Wellness to promote self-reported physical well-being actions in free-living adults who comply with the intervention [3]. The objective of this feasibility study is to address uncertainties regarding the inclusion of accelerometer-based assessment of physical activity within the Fun For Wellness online intervention among free-living adults with obesity in the United States of America.

Four specific aims will be investigated. Aim 1. To determine if accelerometer-based assessment of physical activity can be used within the Fun For Wellness intervention.

Aim 2. To determine if accelerometer-based assessment of physical activity should be used within the Fun For Wellness intervention.

Aim 3. To determine how to implement accelerometer-based assessment of physical activity within the Fun For Wellness intervention.

Aim 4. To provide a preliminary effect size estimate for each direct effect in the conceptual model for the Fun For Wellness online intervention.

Pursuit of these four specific aims is based on a general conceptual framework for feasibility and pilot studies in preparation for a future definitive randomized controlled trial [4-6]. Within this conceptual framework, a randomized pilot trial is a type of a feasibility study and a feasibility study may include a focus on the acceptability of an intervention [4-6].

ELIGIBILITY:
Inclusion Criteria:

Individual is at least 18 years old but not older than 64 years old. Individual has a body mass index (BMI) ≥ 25.00 kg/m2. Individual has access to a technological device (e.g., computer) that can access the online intervention.

Individual is not simultaneously enrolled in another program promoting either well-being or physical activity.

Individual is willing to comply with instructions for physical activity monitoring.

Exclusion Criteria:

Individual is less than 18 years old or older than 64 years old. Individual has a body mass index (BMI) < 25.00. Individual does not have access to a technological device (e.g., computer) that can access the online intervention.

Individual is simultaneously enrolled in another program promoting either well-being or physical activity.

Individual is unwilling to comply with instructions for physical activity monitoring.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
feasibility of accelerometer-based assessment of physical activity (recruitment rate) | Week 0
  The feasibility of accelerometer-based assessment of physical activity will be assessed with recruitment rate. Recruitment rate will be defined as the percentage of patients who select "yes" when asked if they are interested in determining if they are eligible for participation in this study.
feasibility of accelerometer-based assessment of physical activity (eligibility rate) | Week 0
  The feasibility of accelerometer-based assessment of physical activity will be assessed with eligibility rate. Eligibility rate will be defined as the percentage of interested patients who are presented with the informed consent form.
feasibility of accelerometer-based assessment of physical activity (consent rate) | Week 0
  The feasibility of accelerometer-based assessment of physical activity will be assessed with consent rate. Consent rate will be defined as the percentage of eligible patients who consent to participate in this study.
self-efficacy to comply | Week 1
  Self-efficacy to comply will be measured with a single item at Wave 1 (i.e., How confident are you in your current ability to get yourself to complete at least 30 Fun For Wellness post-introductory challenges within the next four weeks?) [11].
  Response to the item will form a self-efficacy to comply score with higher values representing greater self-efficacy to comply. The minimum score will be 0. The maximum score will be 4.
well-being self-efficacy (interpersonal sub-scale) | Week 1
  Well-being self-efficacy will be measured at Wave 1 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 1 to form an interpersonal sub-scale score at Wave 1 with higher values representing greater interpersonal well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (community sub-scale) | Week 1
  Well-being self-efficacy will be measured at Wave 1 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 1 to form a community sub-scale score at Wave 1 with higher values representing greater community well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (occupational sub-scale) | Week 1
  Well-being self-efficacy will be measured at Wave 1 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 1 to form an occupational sub-scale score at Wave 1 with higher values representing greater occupational well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (physical sub-scale) | Week 1
  Well-being self-efficacy will be measured at Wave 1 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 1 to form a physical sub-scale score at Wave 1 with higher values representing greater physical well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (psychological sub-scale) | Week 1
  Well-being self-efficacy will be measured at Wave 1 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 1 to form a psychological sub-scale score at Wave 1 with higher values representing greater psychological well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (economic sub-scale) | Week 1
  Well-being self-efficacy will be measured at Wave 1 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 1 to form an economic sub-scale score at Wave 1 with higher values representing greater economic well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (overall sub-scale) | Week 1
  Well-being self-efficacy will be measured at Wave 1 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the overall sub-scale will be summed at Wave 1 to form an overall sub-scale score at Wave 1 with higher values representing greater overall well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (interpersonal sub-scale) | Week 1
  Well-being actions self-efficacy will be measured at Wave 1 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 1 to form an interpersonal sub-scale score at Wave 1 with higher values representing greater interpersonal well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (community sub-scale) | Week 1
  Well-being actions self-efficacy will be measured at Wave 1 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 1 to form a community sub-scale score at Wave 1 with higher values representing greater community well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (occupational sub-scale) | Week 1
  Well-being actions self-efficacy will be measured at Wave 1 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 1 to form an occupational sub-scale score at Wave 1 with higher values representing greater occupational well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (physical sub-scale) | Week 1
  Well-being actions self-efficacy will be measured at Wave 1 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 1 to form a physical sub-scale score at Wave 1 with higher values representing greater physical well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (psychological sub-scale) | Week 1
  Well-being actions self-efficacy will be measured at Wave 1 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 1 to form a psychological sub-scale score at Wave 1 with higher values representing greater psychological well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (economic sub-scale) | Week 1
  Well-being actions self-efficacy will be measured at Wave 1 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 1 to form an economic sub-scale score at Wave 1 with higher values representing greater economic well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
subjective well-being (interpersonal sub-scale) | Week 1
  Subjective well-being will be measured at Wave 1 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 1 to form an interpersonal sub-scale score at Wave 1 with higher values representing greater interpersonal well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (community sub-scale) | Week 1
  Subjective well-being will be measured at Wave 1 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 1 to form a community sub-scale score at Wave 1 with higher values representing greater interpersonal well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (occupational sub-scale) | Week 1
  Subjective well-being will be measured at Wave 1 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 1 to form an occupational sub-scale score at Wave 1 with higher values representing greater occupational well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (physical sub-scale) | Week 1
  Subjective well-being will be measured at Wave 1 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 1 to form a physical sub-scale score at Wave 1 with higher values representing greater physical well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (psychological sub-scale) | Week 1
  Subjective well-being will be measured at Wave 1 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 1 to form a psychological sub-scale score at Wave 1 with higher values representing greater psychological well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (economic sub-scale) | Week 1
  Subjective well-being will be measured at Wave 1 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 1 to form an economic sub-scale score at Wave 1 with higher values representing greater economic well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (overall sub-scale) | Week 1
  Subjective well-being will be measured at Wave 1 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the overall sub-scale will be summed at Wave 1 to form an overall sub-scale score at Wave 1 with higher values representing greater overall well-being. The minimum score will be 0. The maximum score will be 30.
well-being actions (interpersonal sub-scale) | Week 1
  Well-being actions will be measured at Wave 1 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 1 to form an interpersonal sub-scale score at Wave 1 with higher values representing greater interpersonal well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (community sub-scale) | Week 1
  Well-being actions will be measured at Wave 1 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 1 to form a community sub-scale score at Wave 1 with higher values representing greater community well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (occupational sub-scale) | Week 1
  Well-being actions will be measured at Wave 1 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 1 to form an occupational sub-scale score at Wave 1 with higher values representing greater occupational well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (physical sub-scale) | Week 1
  Well-being actions will be measured at Wave 1 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 1 to form a physical sub-scale score at Wave 1 with higher values representing greater physical well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (psychological sub-scale) | Week 1
  Well-being actions will be measured at Wave 1 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 1 to form a psychological sub-scale score at Wave 1 with higher values representing greater psychological well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (economic sub-scale) | Week 1
  Well-being actions will be measured at Wave 1 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 1 to form an economic sub-scale score at Wave 1 with higher values representing greater psychological well-being actions. The minimum score will be 0. The maximum score will be 12.
physical activity self-efficacy (job-related vigorous sub-scale) | Week 1
  Physical activity self-efficacy will be measured at Wave 1 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the job-related vigorous sub-scale will be summed at Wave 1 to form a job-related vigorous sub-scale score at Wave 1 with higher values representing greater physical activity self-efficacy (job-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (transportation-related vigorous sub-scale) | Week 1
  Physical activity self-efficacy will be measured at Wave 1 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the transportation-related vigorous sub-scale will be summed at Wave 1 to form a transportation-related vigorous sub-scale score at Wave 1 with higher values representing greater physical activity self-efficacy (transportation-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (domestic and gardening-related vigorous sub-scale) | Week 1
  Physical activity self-efficacy will be measured at Wave 1 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the domestic and gardening-related vigorous sub-scale will be summed at Wave 1 to form a domestic and gardening-related vigorous sub-scale score at Wave 1 with higher values representing greater physical activity self-efficacy (domestic and gardening-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (leisure-related vigorous sub-scale) | Week 1
  Physical activity self-efficacy will be measured at Wave 1 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the leisure-related vigorous sub-scale will be summed at Wave 1 to form a leisure-related vigorous sub-scale score at Wave 1 with higher values representing greater physical activity self-efficacy (leisure-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (job-related moderate sub-scale) | Week 1
  Physical activity self-efficacy will be measured at Wave 1 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the job-related moderate sub-scale will be summed at Wave 1 to form a job-related moderate sub-scale score at Wave 1 with higher values representing greater physical activity self-efficacy (job-related moderate). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (transportation-related moderate sub-scale) | Week 1
  Physical activity self-efficacy will be measured at Wave 1 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the transportation-related moderate sub-scale will be summed at Wave 1 to form a transportation-related moderate sub-scale score at Wave 1 with higher values representing greater physical activity self-efficacy (transportation-related moderate). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (domestic and gardening-related moderate sub-scale) | Week 1
  Physical activity self-efficacy will be measured at Wave 1 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the domestic and gardening-related moderate sub-scale will be summed at Wave 1 to form a domestic and gardening-related moderate sub-scale score at Wave 1 with higher values representing greater physical activity self-efficacy (domestic and gardening-related moderate). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (leisure-related moderate sub-scale) | Week 1
  Physical activity self-efficacy will be measured at Wave 1 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the leisure-related moderate sub-scale will be summed at Wave 1 to form a leisure-related moderate sub-scale score at Wave 1 with higher values representing greater physical activity self-efficacy (leisure-related moderate). The minimum score will be 0. The maximum score will be 24.
Self-efficacy to regulate physical activity | Week 1
  Self-efficacy to regulate physical activity will be measured at Wave 1 with the 13-item self-efficacy to regulate physical activity scale [11].
  Responses to the thirteen Likert-scale quantitative items will be summed at Wave 1 to form a a total self-efficacy to regulate physical activity score at Wave 1 with higher values representing greater self-efficacy to regulate physical activity. The minimum score will be 0. The maximum score will be 52.
physical activity (Fitbit Zip) | Week 2
  A commercial-grade (Fitbit Zip) accelerometer will be initialized and attached to an adjustable nylon belt to measure physical activity objectively at Wave 1. Average minutes-per-day of moderate to vigorous physical activity will be determined using the Fitbit application, which uses a proprietary algorithm to estimate fairly active minutes and very active minutes.
physical activity (Actigraph wGT3X-BT) | Week 2
  A research-grade (Actigraph wGT3X-BT) accelerometer will be initialized and attached to an adjustable nylon belt to measure physical activity objectively at Wave 1. Average minutes-per-day of moderate to vigorous physical activity will be calculated based on established cut points (e.g., > 1952 counts per minute).
self-reported physical activity | Week 2
  Self-reported physical activity will be measured at Wave 1 with the long form of the international physical activity questionnaire [9,10]. Average minutes-per-day of moderate to vigorous physical activity will be formed by dividing the sum of the minutes per day (across one week) of minutes-per-day of moderate to vigorous physical activity in the work, transportation, domestic and gardening, and leisure domains by 7 days.
feasibility of accelerometer-based assessment of physical activity (participation rate) | Week 2
  The feasibility of accelerometer-based assessment of physical activity will be assessed with participation rate at Wave 1. Participation rate at Wave 1 will be defined as the percentage of consented patients who provide usable data at Wave 1.
  Usable data will be defined as: (a) a log sheet with a valid start date is submitted, (b) a monitor is worn for at least 4 days (including one weekend day) with at least 10 hours of valid wear time per day, and (c) no evidence of monitor error (e.g., activity counts > 20,000 or lengthy strings of repeated activity counts).
acceptability of accelerometer-based assessment of physical activity (quantitative) | Week 3
  The acceptability of accelerometer-based assessment of physical activity will be assessed at Wave 1 with a modified version of an unnamed questionnaire used in previous research [7,8]. The 11-item acceptability questionnaire used in this study consists of a mix of both Likert-scale quantitative (6) and open-ended qualitative (5) items.
  Responses to the five qualitative items will be content analyzed together at Wave 1 to find conceptual themes at Wave 1 with regard to the acceptability of accelerometer-based assessment of physical activity.
acceptability of accelerometer-based assessment of physical activity (qualitative) | Week 3
  The acceptability of accelerometer-based assessment of physical activity will be assessed at Wave 1 with a modified version of an unnamed questionnaire used in previous research [7,8]. The 11-item acceptability questionnaire used in this study consists of a mix of both Likert-scale quantitative (6) and open-ended qualitative (5) items.
  Responses to the six Likert-scale quantitative items will be summed at Wave 1 to form a total acceptability score at Wave 1 with higher values representing greater acceptability. The minimum total acceptability score at Wave 1 will be 6. The maximum total acceptability score at Wave 1 will be 23.
well-being self-efficacy (interpersonal sub-scale) | Week 7
  Well-being self-efficacy will be measured at Wave 2 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 2 to form an interpersonal sub-scale score at Wave 2 with higher values representing greater interpersonal well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (community sub-scale) | Week 7
  Well-being self-efficacy will be measured at Wave 2 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 2 to form a community sub-scale score at Wave 2 with higher values representing greater community well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (occupational sub-scale) | Week 7
  Well-being self-efficacy will be measured at Wave 2 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 2 to form an occupational sub-scale score at Wave 2 with higher values representing greater occupational well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (physical sub-scale) | Week 7
  Well-being self-efficacy will be measured at Wave 2 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 2 to form a physical sub-scale score at Wave 2 with higher values representing greater physical well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (psychological sub-scale) | Week 7
  Well-being self-efficacy will be measured at Wave 2 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 2 to form a psychological sub-scale score at Wave 2 with higher values representing greater psychological well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (economic sub-scale) | Week 7
  Well-being self-efficacy will be measured at Wave 2 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 2 to form an economic sub-scale score at Wave 2 with higher values representing greater economic well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (overall sub-scale) | Week 7
  Well-being self-efficacy will be measured at Wave 2 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the overall sub-scale will be summed at Wave 2 to form an overall sub-scale score at Wave 2 with higher values representing greater overall well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (interpersonal sub-scale) | Week 7
  Well-being actions self-efficacy will be measured at Wave 2 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 2 to form an interpersonal sub-scale score at Wave 2 with higher values representing greater interpersonal well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (community sub-scale) | Week 7
  Well-being actions self-efficacy will be measured at Wave 2 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 2 to form a community sub-scale score at Wave 2 with higher values representing greater community well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (occupational sub-scale) | Week 7
  Well-being actions self-efficacy will be measured at Wave 2 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 2 to form an occupational sub-scale score at Wave 2 with higher values representing greater occupational well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (physical sub-scale) | Week 7
  Well-being actions self-efficacy will be measured at Wave 2 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 2 to form a physical sub-scale score at Wave 2 with higher values representing greater physical well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (psychological sub-scale) | Week 7
  Well-being actions self-efficacy will be measured at Wave 2 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 2 to form a psychological sub-scale score at Wave 2 with higher values representing greater psychological well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (economic sub-scale) | Week 7
  Well-being actions self-efficacy will be measured at Wave 2 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 2 to form an economic sub-scale score at Wave 2 with higher values representing greater economic well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
subjective well-being (interpersonal sub-scale) | Week 7
  Subjective well-being will be measured at Wave 2 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 2 to form an interpersonal sub-scale score at Wave 2 with higher values representing greater interpersonal well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (community sub-scale) | Week 7
  Subjective well-being will be measured at Wave 2 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 2 to form a community sub-scale score at Wave 2 with higher values representing greater interpersonal well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (occupational sub-scale) | Week 7
  Subjective well-being will be measured at Wave 2 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 2 to form an occupational sub-scale score at Wave 2 with higher values representing greater occupational well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (physical sub-scale) | Week 7
  Subjective well-being will be measured at Wave 2 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 2 to form a physical sub-scale score at Wave 2 with higher values representing greater physical well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (psychological sub-scale) | Week 7
  Subjective well-being will be measured at Wave 2 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 2 to form a psychological sub-scale score at Wave 2 with higher values representing greater psychological well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (economic sub-scale) | Week 7
  Subjective well-being will be measured at Wave 2 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 2 to form an economic sub-scale score at Wave 2 with higher values representing greater economic well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (overall sub-scale) | Week 7
  Subjective well-being will be measured at Wave 2 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the overall sub-scale will be summed at Wave 2 to form an overall sub-scale score at Wave 2 with higher values representing greater overall well-being. The minimum score will be 0. The maximum score will be 30.
well-being actions (interpersonal sub-scale) | Week 7
  Well-being actions will be measured at Wave 2 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 2 to form an interpersonal sub-scale score at Wave 2 with higher values representing greater interpersonal well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (community sub-scale) | Week 7
  Well-being actions will be measured at Wave 2 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 2 to form a community sub-scale score at Wave 2 with higher values representing greater community well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (occupational sub-scale) | Week 7
  Well-being actions will be measured at Wave 2 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 2 to form an occupational sub-scale score at Wave 2 with higher values representing greater occupational well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (physical sub-scale) | Week 7
  Well-being actions will be measured at Wave 2 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 2 to form a physical sub-scale score at Wave 2 with higher values representing greater physical well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (psychological sub-scale) | Week 7
  Well-being actions will be measured at Wave 2 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 2 to form a psychological sub-scale score at Wave 2 with higher values representing greater psychological well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (economic sub-scale) | Week 7
  Well-being actions will be measured at Wave 2 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 2 to form an economic sub-scale score at Wave 2 with higher values representing greater psychological well-being actions. The minimum score will be 0. The maximum score will be 12.
physical activity self-efficacy (job-related vigorous sub-scale) | Week 7
  Physical activity self-efficacy will be measured at Wave 2 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the job-related vigorous sub-scale will be summed at Wave 2 to form a job-related vigorous sub-scale score at Wave 2 with higher values representing greater physical activity self-efficacy (job-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (transportation-related vigorous sub-scale) | Week 7
  Physical activity self-efficacy will be measured at Wave 2 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the transportation-related vigorous sub-scale will be summed at Wave 2 to form a transportation-related vigorous sub-scale score at Wave 2 with higher values representing greater physical activity self-efficacy (transportation-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (domestic and gardening-related vigorous sub-scale) | Week 7
  Physical activity self-efficacy will be measured at Wave 2 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the domestic and gardening-related vigorous sub-scale will be summed at Wave 2 to form a domestic and gardening-related vigorous sub-scale score at Wave 2 with higher values representing greater physical activity self-efficacy (domestic and gardening-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (leisure-related vigorous sub-scale) | Week 7
  Physical activity self-efficacy will be measured at Wave 2 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the leisure-related vigorous sub-scale will be summed at Wave 2 to form a leisure-related vigorous sub-scale score at Wave 2 with higher values representing greater physical activity self-efficacy (leisure-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (job-related moderate sub-scale) | Week 7
  Physical activity self-efficacy will be measured at Wave 2 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the job-related moderate sub-scale will be summed at Wave 2 to form a job-related moderate sub-scale score at Wave 2 with higher values representing greater physical activity self-efficacy (job-related moderate). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (transportation-related moderate sub-scale) | Week 7
  Physical activity self-efficacy will be measured at Wave 2 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the transportation-related moderate sub-scale will be summed at Wave 2 to form a transportation-related moderate sub-scale score at Wave 2 with higher values representing greater physical activity self-efficacy (transportation-related moderate). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (domestic and gardening-related moderate sub-scale) | Week 7
  Physical activity self-efficacy will be measured at Wave 2 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the domestic and gardening-related moderate sub-scale will be summed at Wave 2 to form a domestic and gardening-related moderate sub-scale score at Wave 2 with higher values representing greater physical activity self-efficacy (domestic and gardening-related moderate). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (leisure-related moderate sub-scale) | Week 7
  Physical activity self-efficacy will be measured at Wave 2 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the leisure-related moderate sub-scale will be summed at Wave 2 to form a leisure-related moderate sub-scale score at Wave 2 with higher values representing greater physical activity self-efficacy (leisure-related moderate). The minimum score will be 0. The maximum score will be 24.
Self-efficacy to regulate physical activity | Week 7
  Self-efficacy to regulate physical activity will be measured at Wave 2 with the 13-item self-efficacy to regulate physical activity scale [11].
  Responses to the thirteen Likert-scale quantitative items will be summed at Wave 2 to form a a total self-efficacy to regulate physical activity score at Wave 2 with higher values representing greater self-efficacy to regulate physical activity. The minimum score will be 0. The maximum score will be 52.
physical activity (Actigraph wGT3X-BT) | Week 8
  A research-grade (Actigraph wGT3X-BT) accelerometer will be initialized and attached to an adjustable nylon belt to measure physical activity objectively at Wave 2. Average minutes-per-day of moderate to vigorous physical activity will be calculated based on established cut points (e.g., > 1952 counts per minute).
self-reported physical activity | Week 8
  Self-reported physical activity will be measured at Wave 2 with the long form of the international physical activity questionnaire [9,10]. Average minutes-per-day of moderate to vigorous physical activity will be formed by dividing the sum of the minutes per day (across one week) of minutes-per-day of moderate to vigorous physical activity in the work, transportation, domestic and gardening, and leisure domains by 7 days.
physical activity (Fitbit Zip) | Week 8
  A commercial-grade (Fitbit Zip) accelerometer will be initialized and attached to an adjustable nylon belt to measure physical activity objectively at Wave 2. Average minutes-per-day of moderate to vigorous physical activity will be determined using the Fitbit application, which uses a proprietary algorithm to estimate fairly active minutes and very active minutes.
feasibility of accelerometer-based assessment of physical activity (participation rate) | Week 8
  The feasibility of accelerometer-based assessment of physical activity will be assessed with participation rate at Wave 2. Participation rate at Wave 2 will be defined as the percentage of consented patients who provide usable data at Wave 2.
  Usable data will be defined as: (a) a log sheet with a valid start date is submitted, (b) a monitor is worn for at least 4 days (including one weekend day) with at least 10 hours of valid wear time per day, and (c) no evidence of monitor error (e.g., activity counts > 20,000 or lengthy strings of repeated activity counts).
feasibility of accelerometer-based assessment of physical activity (retention rate) | Week 8
  The feasibility of accelerometer-based assessment of physical activity will be assessed with retention rate at Wave 2. Retention rate at Wave 2 will be defined as the percentage of consented patients who provide usable data at Wave 1 and Wave 2.
  Usable data will be defined as: (a) a log sheet with a valid start date is submitted, (b) a monitor is worn for at least 4 days (including one weekend day) with at least 10 hours of valid wear time per day, and (c) no evidence of monitor error (e.g., activity counts > 20,000 or lengthy strings of repeated activity counts).
acceptability of accelerometer-based assessment of physical activity (quantitative) | Week 9
  The acceptability of accelerometer-based assessment of physical activity will be assessed at Wave 2 with a modified version of an unnamed questionnaire used in previous research [7,8]. The 11-item acceptability questionnaire used in this study consists of a mix of both Likert-scale quantitative (6) and open-ended qualitative (5) items.
  Responses to the six Likert-scale quantitative items will be summed at Wave 2 to form a total acceptability score at Wave 2 with higher values representing greater acceptability. The minimum total acceptability score at Wave 2 will be 6. The maximum total acceptability score at Wave 2 will be 23.
acceptability of accelerometer-based assessment of physical activity (qualitative) | Week 9
  The acceptability of accelerometer-based assessment of physical activity will be assessed at Wave 2 with a modified version of an unnamed questionnaire used in previous research [7,8]. The 11-item acceptability questionnaire used in this study consists of a mix of both Likert-scale quantitative (6) and open-ended qualitative (5) items.
  Responses to the five qualitative items will be content analyzed together at Wave 2 to find conceptual themes at Wave 2 with regard to the acceptability of accelerometer-based assessment of physical activity.
well-being self-efficacy (interpersonal sub-scale) | Week 11
  Well-being self-efficacy will be measured at Wave 3 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 3 to form an interpersonal sub-scale score at Wave 2 with higher values representing greater interpersonal well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (community sub-scale) | Week 11
  Well-being self-efficacy will be measured at Wave 3 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 3 to form a community sub-scale score at Wave 3 with higher values representing greater community well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (occupational sub-scale) | Week 11
  Well-being self-efficacy will be measured at Wave 3 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 3 to form an occupational sub-scale score at Wave 3 with higher values representing greater occupational well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (physical sub-scale) | Week 11
  Well-being self-efficacy will be measured at Wave 3 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 3 to form a physical sub-scale score at Wave 3 with higher values representing greater physical well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (psychological sub-scale) | Week 11
  Well-being self-efficacy will be measured at Wave 3 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 3 to form a psychological sub-scale score at Wave 3 with higher values representing greater psychological well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (economic sub-scale) | Week 11
  Well-being self-efficacy will be measured at Wave 3 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 3 to form an economic sub-scale score at Wave 3 with higher values representing greater economic well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being self-efficacy (overall sub-scale) | Week 11
  Well-being self-efficacy will be measured at Wave 3 with the 21-item well-being self-efficacy scale [1,11].
  Responses to the three Likert-scale quantitative items intended to measure the overall sub-scale will be summed at Wave 3 to form an overall sub-scale score at Wave 3 with higher values representing greater overall well-being self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (interpersonal sub-scale) | Week 11
  Well-being actions self-efficacy will be measured at Wave 3 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 3 to form an interpersonal sub-scale score at Wave 3 with higher values representing greater interpersonal well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (community sub-scale) | Week 11
  Well-being actions self-efficacy will be measured at Wave 3 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 3 to form a community sub-scale score at Wave 3 with higher values representing greater community well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (occupational sub-scale) | Week 11
  Well-being actions self-efficacy will be measured at Wave 3 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 3 to form an occupational sub-scale score at Wave 3 with higher values representing greater occupational well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (physical sub-scale) | Week 11
  Well-being actions self-efficacy will be measured at Wave 3 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 3 to form a physical sub-scale score at Wave 3 with higher values representing greater physical well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (psychological sub-scale) | Week 11
  Well-being actions self-efficacy will be measured at Wave 3 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 3 to form a psychological sub-scale score at Wave 3 with higher values representing greater psychological well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
well-being actions self-efficacy (economic sub-scale) | Week 11
  Well-being actions self-efficacy will be measured at Wave 3 with the 18-item well-being actions self-efficacy scale [11].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 3 to form an economic sub-scale score at Wave 3 with higher values representing greater economic well-being actions self efficacy. The minimum score will be 0. The maximum score will be 12.
subjective well-being (interpersonal sub-scale) | Week 11
  Subjective well-being will be measured at Wave 3 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 3 to form an interpersonal sub-scale score at Wave 3 with higher values representing greater interpersonal well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (community sub-scale) | Week 11
  Subjective well-being will be measured at Wave 3 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 3 to form a community sub-scale score at Wave 3 with higher values representing greater interpersonal well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (occupational sub-scale) | Week 11
  Subjective well-being will be measured at Wave 3 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 3 to form an occupational sub-scale score at Wave 3 with higher values representing greater occupational well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (physical sub-scale) | Week 11
  Subjective well-being will be measured at Wave 3 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 3 to form a physical sub-scale score at Wave 3 with higher values representing greater physical well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (psychological sub-scale) | Week 11
  Subjective well-being will be measured at Wave 3 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 3 to form a psychological sub-scale score at Wave 3 with higher values representing greater psychological well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (economic sub-scale) | Week 11
  Subjective well-being will be measured at Wave 3 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 3 to form an economic sub-scale score at Wave 3 with higher values representing greater economic well-being. The minimum score will be 0. The maximum score will be 30.
subjective well-being (overall sub-scale) | Week 11
  Subjective well-being will be measured at Wave 3 with the 21-item I COPPE scale [12].
  Responses to the three Likert-scale quantitative items intended to measure the overall sub-scale will be summed at Wave 3 to form an overall sub-scale score at Wave 3 with higher values representing greater overall well-being. The minimum score will be 0. The maximum score will be 30.
well-being actions (interpersonal sub-scale) | Week 11
  Well-being actions will be measured at Wave 3 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the interpersonal sub-scale will be summed at Wave 3 to form an interpersonal sub-scale score at Wave 3 with higher values representing greater interpersonal well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (community sub-scale) | Week 11
  Well-being actions will be measured at Wave 3 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the community sub-scale will be summed at Wave 3 to form a community sub-scale score at Wave 3 with higher values representing greater community well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (occupational sub-scale) | Week 11
  Well-being actions will be measured at Wave 3 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the occupational sub-scale will be summed at Wave 3 to form an occupational sub-scale score at Wave 3 with higher values representing greater occupational well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (physical sub-scale) | Week 11
  Well-being actions will be measured at Wave 3 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the physical sub-scale will be summed at Wave 3 to form a physical sub-scale score at Wave 3 with higher values representing greater physical well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (psychological sub-scale) | Week 11
  Well-being actions will be measured at Wave 3 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the psychological sub-scale will be summed at Wave 3 to form a psychological sub-scale score at Wave 3 with higher values representing greater psychological well-being actions. The minimum score will be 0. The maximum score will be 12.
well-being actions (economic sub-scale) | Week 11
  Well-being actions will be measured at Wave 3 with the 18-item I COPPE actions scale [13].
  Responses to the three Likert-scale quantitative items intended to measure the economic sub-scale will be summed at Wave 3 to form an economic sub-scale score at Wave 3 with higher values representing greater psychological well-being actions. The minimum score will be 0. The maximum score will be 12.
physical activity self-efficacy (job-related vigorous sub-scale) | Week 11
  Physical activity self-efficacy will be measured at Wave 3 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the job-related vigorous sub-scale will be summed at Wave 3 to form a job-related vigorous sub-scale score at Wave 3 with higher values representing greater physical activity self-efficacy (job-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (domestic and gardening-related vigorous sub-scale) | Week 11
  Physical activity self-efficacy will be measured at Wave 3 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the domestic and gardening-related vigorous sub-scale will be summed at Wave 3 to form a domestic and gardening-related vigorous sub-scale score at Wave 3 with higher values representing greater physical activity self-efficacy (domestic and gardening-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (transportation-related vigorous sub-scale) | Week 11
  Physical activity self-efficacy will be measured at Wave 3 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the transportation-related vigorous sub-scale will be summed at Wave 3 to form a transportation-related vigorous sub-scale score at Wave 3 with higher values representing greater physical activity self-efficacy (transportation-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (leisure-related vigorous sub-scale) | Week 11
  Physical activity self-efficacy will be measured at Wave 3 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the leisure-related vigorous sub-scale will be summed at Wave 3 to form a leisure-related vigorous sub-scale score at Wave 3 with higher values representing greater physical activity self-efficacy (leisure-related vigorous). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (job-related moderate sub-scale) | Week 11
  Physical activity self-efficacy will be measured at Wave 3 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the job-related moderate sub-scale will be summed at Wave 3 to form a job-related moderate sub-scale score at Wave 3 with higher values representing greater physical activity self-efficacy (job-related moderate). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (transportation-related moderate sub-scale) | Week 11
  Physical activity self-efficacy will be measured at Wave 3 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the transportation-related moderate sub-scale will be summed at Wave 3 to form a transportation-related moderate sub-scale score at Wave 3 with higher values representing greater physical activity self-efficacy (transportation-related moderate). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (domestic and gardening-related moderate sub-scale) | Week 11
  Physical activity self-efficacy will be measured at Wave 3 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the domestic and gardening-related moderate sub-scale will be summed at Wave 3 to form a domestic and gardening-related moderate sub-scale score at Wave 3 with higher values representing greater physical activity self-efficacy (domestic and gardening-related moderate). The minimum score will be 0. The maximum score will be 24.
physical activity self-efficacy (leisure-related moderate sub-scale) | Week 11
  Physical activity self-efficacy will be measured at Wave 3 with the 48-item physical activity self-efficacy scale [11].
  Responses to the six Likert-scale quantitative items intended to measure the leisure-related moderate sub-scale will be summed at Wave 3 to form a leisure-related moderate sub-scale score at Wave 3 with higher values representing greater physical activity self-efficacy (leisure-related moderate). The minimum score will be 0. The maximum score will be 24.
Self-efficacy to regulate physical activity | Week 11
  Self-efficacy to regulate physical activity will be measured at Wave 3 with the 13-item self-efficacy to regulate physical activity scale [11].
  Responses to the thirteen Likert-scale quantitative items will be summed at Wave 3 to form a a total self-efficacy to regulate physical activity score at Wave 3 with higher values representing greater self-efficacy to regulate physical activity. The minimum score will be 0. The maximum score will be 52.
physical activity (Fitbit Zip) | Week 12
  A commercial-grade (Fitbit Zip) accelerometer will be initialized and attached to an adjustable nylon belt to measure physical activity objectively at Wave 3. Average minutes-per-day of moderate to vigorous physical activity will be determined using the Fitbit application, which uses a proprietary algorithm to estimate fairly active minutes and very active minutes.
physical activity (Actigraph wGT3X-BT) | Week 12
  A research-grade (Actigraph wGT3X-BT) accelerometer will be initialized and attached to an adjustable nylon belt to measure physical activity objectively at Wave 3. Average minutes-per-day of moderate to vigorous physical activity will be calculated based on established cut points (e.g., > 1952 counts per minute).
self-reported physical activity | Week 12
  Self-reported physical activity will be measured at Wave 3 with the long form of the international physical activity questionnaire [9,10]. Average minutes-per-day of moderate to vigorous physical activity will be formed by dividing the sum of the minutes per day (across one week) of minutes-per-day of moderate to vigorous physical activity in the work, transportation, domestic and gardening, and leisure domains by 7 days.
feasibility of accelerometer-based assessment of physical activity (participation rate) | Week 12
  The feasibility of accelerometer-based assessment of physical activity will be assessed with participation rate at Wave 3. Participation rate at Wave 1 will be defined as the percentage of consented patients who provide usable data at Wave 3.
  Usable data will be defined as: (a) a log sheet with a valid start date is submitted, (b) a monitor is worn for at least 4 days (including one weekend day) with at least 10 hours of valid wear time per day, and (c) no evidence of monitor error (e.g., activity counts > 20,000 or lengthy strings of repeated activity counts).
feasibility of accelerometer-based assessment of physical activity (retention rate) | Week 12
  The feasibility of accelerometer-based assessment of physical activity will be assessed with retention rate at Wave 3. Retention rate at Wave 3 will be defined as the percentage of consented patients who provide usable data at Wave 1, Wave 2, and Wave 3.
  Usable data will be defined as: (a) a log sheet with a valid start date is submitted, (b) a monitor is worn for at least 4 days (including one weekend day) with at least 10 hours of valid wear time per day, and (c) no evidence of monitor error (e.g., activity counts > 20,000 or lengthy strings of repeated activity counts).
acceptability of accelerometer-based assessment of physical activity (quantitative) | Week 13
  The acceptability of accelerometer-based assessment of physical activity will be assessed at Wave 3 with a modified version of an unnamed questionnaire used in previous research [7,8]. The 11-item acceptability questionnaire used in this study consists of a mix of both Likert-scale quantitative (6) and open-ended qualitative (5) items.
  Responses to the six Likert-scale quantitative items will be summed at Wave 3 to form a total acceptability score at Wave 3 with higher values representing greater acceptability. The minimum total acceptability score at Wave 3 will be 6. The maximum total acceptability score at Wave 3 will be 23.
acceptability of accelerometer-based assessment of physical activity (qualitative) | Week 13
  The acceptability of accelerometer-based assessment of physical activity will be assessed at Wave 3 with a modified version of an unnamed questionnaire used in previous research [7,8]. The 11-item acceptability questionnaire used in this study consists of a mix of both Likert-scale quantitative (6) and open-ended qualitative (5) items.
  Responses to the five qualitative items will be content analyzed together at Wave 3 to find conceptual themes at Wave 3 with regard to the acceptability of accelerometer-based assessment of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas D Myers, Ph.D., Principal Investigator — Michigan State University; Isaac Prilleltensky, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Sparrow Health System Bariatric Services, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myers ND, Prilleltensky I, Prilleltensky O, McMahon A, Dietz S, Rubenstein CL. Efficacy of the Fun For Wellness Online Intervention to Promote Multidimensional Well-Being: a Randomized Controlled Trial. Prev Sci. 2017 Nov;18(8):984-994. doi: 10.1007/s11121-017-0779-z. PMID 28303422
- [Background] Bandura A. Self-efficacy: the exercise of control. New York: Freeman; 1997.
- [Background] Myers ND, Dietz S, Prilleltensky I, Prilleltensky O, McMahon A, Rubenstein CL, Lee S. Efficacy of the Fun For Wellness Online Intervention to Promote Well-Being Actions: A Secondary Data Analysis. Games Health J. 2018 Aug;7(4):225-239. doi: 10.1089/g4h.2017.0132. Epub 2018 Apr 30. PMID 29708773
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Thabane L, Hopewell S, Lancaster GA, Bond CM, Coleman CL, Campbell MJ, Eldridge SM. Erratum to: Methods and processes for development of a CONSORT extension for reporting pilot randomized controlled trials. Pilot Feasibility Stud. 2016 Jul 19;2:35. doi: 10.1186/s40814-016-0078-7. eCollection 2016. PMID 27976755
- [Background] Tully MA, McBride C, Heron L, Hunter RF. The validation of Fibit Zip physical activity monitor as a measure of free-living physical activity. BMC Res Notes. 2014 Dec 23;7:952. doi: 10.1186/1756-0500-7-952. PMID 25539733
- [Background] Hale LA, Pal J, Becker I. Measuring free-living physical activity in adults with and without neurologic dysfunction with a triaxial accelerometer. Arch Phys Med Rehabil. 2008 Sep;89(9):1765-71. doi: 10.1016/j.apmr.2008.02.027. PMID 18760161
- [Background] Ainsworth BE, Bassett DR Jr, Strath SJ, Swartz AM, O'Brien WL, Thompson RW, Jones DA, Macera CA, Kimsey CD. Comparison of three methods for measuring the time spent in physical activity. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S457-64. doi: 10.1097/00005768-200009001-00004. PMID 10993415
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] ClinicalTrials.gov: Well-Being and Physical Activity Study. https://clinicaltrials.gov/ct2/show/NCT 03194854 Accessed 9 January 2019.
- [Background] Prilleltensky I, Dietz S, Prilleltensky O, Myers ND, Rubenstein CL, Jin Y, et al. Assessing multidimensional well-being: development and validation of the I COPPE scale. J Community Psychol. 2015;43:199-226.
- [Background] Rubenstein CL. Assessing actions and feelings related to multidimensional well-being: validation of the I COPPE actions and feelings scales. 2017. https://scholarlyrepository.miami.edu/oa_dissertations/1942. Accessed 1 July 2018.
- [Derived] Myers ND, Lee S, Bateman AG, Prilleltensky I, Clevenger KA, Pfeiffer KA, Dietz S, Prilleltensky O, McMahon A, Brincks AM. Accelerometer-based assessment of physical activity within the Fun For Wellness online behavioral intervention: protocol for a feasibility study. Pilot Feasibility Stud. 2019 May 31;5:73. doi: 10.1186/s40814-019-0455-0. eCollection 2019. PMID 31164990